CLINICAL TRIAL: NCT02930967
Title: A Safety and Efficacy Study of Chimeric Switch Receptor Modified T Cells in Patients With Recurrent or Metastatic Malignant Tumors
Brief Title: Chimeric Switch Receptor Modified T Cells for Patients With PD-L1+ Recurrent or Metastatic Malignant Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Meitan General Hospital (Other)
Collaborators: Marino Biotechnology Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jinwen Sun, Director of Department of General Surgery and Surgical Oncology, China Meitan General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K16-3
Record Dates: First submitted 2016-10-10; First posted 2016-10-12 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Recurrent PD-L1+ Malignant Tumors; Metastatic PD-L1+ Malignant Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CSR T cells (Experimental): A dose escalation clinical study aimed to assess the safety and efficacy of CSR T cells in patients with PD-L1 positive tumors.
  CSR T dosage ranging from: 5×10^4 /kg to 1×10^7 /kg will be tested.
  Interventions: Biological: autologous CSR T

INTERVENTIONS:
Biological: autologous CSR T — Patients will be received a three-day regimen of chemotherapy consisting of cyclophosphamide aimed to deplete the lymphocytes. 1 to 4 days after lymphodepletion, a prescribed dose of CSR T cells will be intravenously infused to patient in a three-day split-dose regimen (day0,10%; day1, 30%; day2, 60%).

SUMMARY:
A Chimeric Switch Receptor, which was constructed by fusing the PD1 extracellular ligand binding domain to the CD28 intracellular costimulatory domain, was designed to target PD-L 1 positive tumors . In this single-arm, open-label, one center, dose escalation clinical study, the main purpose is to determine the safety and efficacy of infusion of autologous Chimeric Switch Receptor modified T cells (CSR T) in adult patients with PD-L1 positive, recurrent or metastatic malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with PD-L1 positive, recurrent or metastatic malignant tumors , including but not limited to pancreatic cancer, renal cancer, colorectal cancer, lymphoma, breast cancer and lung cancer;
2. measurable tumors by RECIST1.1 standard;
3. patients are 18 to 70 years old;
4. life expectancy > 3months;
5. KPS ≥70;
6. satisfactory major organ functions: adequate heart function with LVEF≥50%; no obvious abnormities in ECG; pulse oximetry ≥ 90%; cockcroft-gault creatinine clearance≥40 ml/min; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3ULN; Bilirubin ≤2.0 mg/dl ;
7. Blood: Hgb ≥ 80 g/L, ANC ≥ 1×10^9/L, PLT ≥ 50×10^9/L;
8. women of reproductive potential must have a negative pregnancy test. Male and female of reproductive potential must agree to use birth control during the study and one year post study.

Exclusion Criteria:

1. patients with a prior history of autoimmune disease or other diseases who need long-term use of systemic hormone drug or immunosuppressive therapy
2. active infection.
3. HIV positive.
4. active hepatitis B virus infection or hepatitis C virus infection.
5. currently enrolled in other study.
6. patients, in the opinion of investigators, may not be eligible or are not able to comply with the study.
7. patients with allergic disease, or are allergic to T cell products or other biological agents used in the study.
8. patients whose tumors have metastasized to bone, or have clinical signs of bone metastasis, such as bone and joint pain.
9. patients with brain metastasis, or have clinical signs of brain metastasis, such as loss of self-consciousness.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Safety as assessed by incidents of treatment related adverse events as assessed by CTCAE V4.0. | 2 years
  safety of infusion of autologous CSR T cells with cyclophosphamide as lymphodepleting chemotherapy

SECONDARY OUTCOMES:
treatment response rate of CSR T cell infusion | 4 weeks
  defined as the proportion of patients who achieved complete remission (CR), partial remission (PR), stable disease (SD), or progressive disease (PD).
overall survival rate | 2 years
progression-free survival | 6 months
proliferation of CSR T cells in patients | 2 years
Persistence of CSR T cells in patients | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jinwen Sun, MD, Principal Investigator — China Meitan General Hospital
Locations (1):
- China Meitan General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided